CLINICAL TRIAL: NCT00586573
Title: An Open-Label Pilot Study of Namenda (Memantine Hydrochloride) in Adult Subjects With Attention Deficit Hyperactivity Disorder (ADHD) and ADHD NOS
Brief Title: Open-Label Pilot Study of Namenda in Adult Subjects With ADHD and ADHD NOS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Paul Hammerness, MD, Assistant Professor Psychiatry, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-P-000067
Record Dates: First submitted 2007-12-28; First posted 2008-01-04 (Estimated); Results first posted 2012-06-07 (Estimated); Last update posted 2012-06-07 (Estimated); Status verified 2012-05

CONDITIONS: ADHD
Keywords: ADHD; Namenda
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Memantine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Namenda (Experimental)
  Interventions: Drug: memantine hydrochloride

INTERVENTIONS:
Drug: memantine hydrochloride — tablet, 5-20 mg, twice daily, by mouth, 12 weeks
  Other Names: Namenda

SUMMARY:
The primary objective of the study is to assess the efficacy and tolerability of a 12-week trial of memantine hydrochloride administered twice daily in 20 adults (ages 18-55) with ADHD and ADHD NOS. Improvement will be defined as: 1) changes from baseline on the investigator-rated DSM-IV based ADHD Rating Scale; 2) changes from baseline in a questionnaire aimed at assessing executive functions (BRIEF); and 3) changes from screening in a computerized neuropsychological battery (CANTAB). We hypothesize that memantine hydrochloride will be associated with improving ADHD symptoms and associated deficits in executive functions. We also expect that memantine will be well-tolerated with predictable adverse events.

DETAILED DESCRIPTION:
Memantine (Namenda) is a low-affinity N-methyl-D-aspartate (NMDA) receptor antagonist believed to work by blocking prolonged low-level activation of the NMDA receptor and resultant neuronal damage caused by abnormal glutamatergic activity, yet also allowing normal physiological activity of the NMDA channel. Memantine (Namenda) was approved by the U.S. Food and Drug Administration in 2003 for the treatment of moderate to severe Alzheimer's disease. Memantine improves or delays the decline in cognition (attention, language, visuo-spatial ability), as well as functional and behavioral symptoms in adults with moderate Alzheimer's disease.

Although the efficacy and safety of memantine has not been tested in people with ADHD, the spectrum of disorders possibly amenable to NMDA receptor antagonist treatment may include ADHD and associated executive function deficits (EFDs). To this end, we are proposing an open-label pilot study of memantine in adult subjects with ADHD and ADHD Not Otherwise Specified (NOS).

This will be a 12-week, open-label pilot study to assess the efficacy and tolerability of memantine hydrochloride (Namenda) administered to 20 adults 18-55 years of age with ADHD and ADHD NOS. All subjects that enter the study will undergo standard screening and diagnostic procedures. After obtaining written informed consent from the subject, the diagnosis of ADHD will be established through clinical evaluation by an expert clinician. Only consenting subjects satisfying inclusion and exclusion criteria will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female outpatients 18-55 years of age
2. Subjects with the diagnosis of Attention Deficit Hyperactivity Disorder (ADHD), by DSM-IV or ADHD NOS (late onset; >7 years), as manifested in clinical evaluation and confirmed by structured interview.
3. Subjects must score at least 14 on inattentive symptom questions on the DSM-IV based ADHD Rating Scale.
4. Subjects who have an ADHD specific CGI Severity score of 4 or more (> moderately impaired).

Exclusion Criteria:

1. Subjects with a medical condition or treatment that will either jeopardize subject safety or affect the scientific merit of the study, including:
2. History of Renal or Hepatic Impairment.
3. Organic brain disorders.
4. History of Seizure disorder.
5. Any clinically unstable psychiatric conditions including the following: psychosis, suicidality, bipolar disorder, current substance use disorders (alcohol or drugs) or current tic disorder.
6. Mental retardation (IQ <75).
7. Pregnant or nursing females.
8. Known hypersensitivity to memantine.
9. Any current psychotropic treatment, with the exception of stable regimen of SSRIs.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2007-03; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Hammerness, MD, Principal Investigator — MGH
Locations (1):
- Massachusetts General Hospital, Cambridge, Massachusetts, United States

REFERENCES:
- See also: Related Info — http://massgeneral.org/pediatricpsych/home.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Memantine: 5-20 mg, twice daily, by mouth, 12 weeks
Period: Overall Study
Arm/Group | Memantine
Started | 34
Completed | 28
Not Completed | 6

BASELINE CHARACTERISTICS:
Arm/Group | Memantine
Number analyzed (Participants) | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 34
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 41.8 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 25

OUTCOME MEASURES:

1. Primary Outcome: DSM-IV ADHD Rating Scale (AISRS) Score Change
Description: AISRS used to assess 18 individual criteria symptoms of ADHD in DSM-IV on a severity grid (0=not present, 3=severe; minimum score=0, maximum score=54). This is a composite score assessing both inattention and hyperactivity, which are not assessed individually in this scale.
  Score change from baseline.
Time Frame: Endpoint, following 12 weeks Memantine Monotherapy
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Memantine
Number analyzed (Participants) | 34
Units on a scale
  Total Symptoms | -17.5 [-22.3 to -12.6]
  Inattentive Symptoms | -10.6 [-13.7 to -7.5]
  Hyperactive Symptoms | -6.9 [-9.0 to -4.7]

ADVERSE EVENTS:
Arm/Group | Memantine
Serious Adverse Events (participants affected / at risk) | 0/34
Other Adverse Events (participants affected / at risk) | 34/34
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Memantine (N=34)
Dizzy/Lightheaded (General disorders) | 8 (10)
Gastrointestinal (Gastrointestinal disorders) | 6 (13)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 6 (13)
Headaches (General disorders) | 5 (12)
Sedation (General disorders) | 4 (7)
Decreased Energy (General disorders) | 3 (4)
Anxiety (Psychiatric disorders) | 2 (2)
Cold/infection/allergy (Infections and infestations) | 2 (11)
Hearing change (Ear and labyrinth disorders) | 1 (1)
Impaired concentration (General disorders) | 2 (7)
Insomnia (General disorders) | 2 (6)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Change in sexual function (Reproductive system and breast disorders) | 1 (2)
Decreased appetite (Gastrointestinal disorders) | 1 (1)
Increased energy (General disorders) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 1 (3)
Mucosal dryness (General disorders) | 1 (4)
Palpitation (Cardiac disorders) | 1 (1)
Tense/jittery (General disorders) | 1 (5)
Vision/ocular (Eye disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No